CLINICAL TRIAL: NCT06988644
Title: Prospective Study Aimed at Evaluating the Effect of a Counseling Consultation in the Workplace for Smoker Employees in a Mental Health Establishment
Brief Title: Impact of a Counseling Consultation in the Workplace for Smoker Health Professionals
Acronym: PSYTaB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier Mutualiste de Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PSYTaB; 2024-A01826-41 (Other: ANSM)
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation; Smoking consultation; carbon monoxyde measurement
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: * Interventional study
  * Prospective
  * Non-randomised
  * Comparative with historical cohort
  * Monocentric
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- consultation tabacco (Experimental): At the first T0 consultation, the tobacco nurse :
  * Carries out a monoxyde carbon measurement, In order to assess the patient's smoking profile and find out their degree of nicotine dependency, what might be holding them back from quitting, what might be motivating them, their psychological state, their fears and their medical history.
  * Define a programme for smoking cessation : the planned date for cessation, the treatment chosen, any additional specific therapy or consultations, and the date of the next appointments.
  During the 6-month follow-up sessions, the nurse assesses the patient's mood and anxiety, with a view to adapting the treatment if necessary.
  At the final consultation at T12 months, the nurse assesses the patient's withdrawal and the effect of the follow-up tobacco consultations.
  Interventions: Diagnostic Test: exhaled carbon monoxyde measurement

INTERVENTIONS:
Diagnostic Test: exhaled carbon monoxyde measurement — At the initial tobacco consultation: measurement of exhaled carbon monoxyde. At the tobaccology consultation at 12 months, measurement of the cessation rate: no tobacco smoked in the last 7 days (self-reported), confirmed by a measurement of exhaled carbon monoxyde < 9 ppm.

SUMMARY:
Smoking is still a major cause of premature death in France (75,000 deaths a year). Health professionals also seem to be affected by smoking, but few studies have been carried out on this population of smokers. While having a job can be protective, certain working conditions are at risk: night shifts, stress, physical strain, burnout... In 2010, 23% of nurses and 40% of nursing auxiliaries were smokers. More recently, a study of 10,000 health professionals in a French health establishment in 2022 revealed a rate of 32% among nursing auxiliaries.

Data on smoking among health professionals is still scarce. Yet they seem essential, given that smoking among healthcare professionals seems to be an obstacle to dealing with patients' consumption and contributes to the erroneous representations that persist in psychiatry more than elsewhere, such as: "smoking with a patient makes an alliance with them", "smoking is a way of reducing psychological tension", "patients have other problems to deal with", "it won't work because they've been smoking for years". Smoking in mental health facilities is high among both patients and professionals.

Investigators now know that smoking has an impact on mood disorders and sleep. It aggravates all somatic and psychological pathologies and predisposes people to more diabetes, chronic bronchitis, cardiovascular disease, cancer, etc. It also interacts with many drugs.

Smoking screening and cessation assistance have become an indicator of quality somatic care in mental health institutions.

Investigators hypothesise that a consultation in the workplace can help employees to change their smoking habits.

The aims of this study are to assess the effect of a workplace smoking clinic on smokers employed in a mental health institution, and to describe their smoking habits and profiles according to occupational category, with a view to implementing appropriate preventive and treatment measures.

DETAILED DESCRIPTION:
Smoking is still a major cause of premature death in France (75,000 deaths a year). Healthcare professionals also seem to be affected by smoking, and few studies have been carried out on this population of smokers.

In 2010, 23% of nurses and 40% of nursing auxiliaries in France said they smoked every day. In a more recent study on parisian hospitals, the prevalence of daily smoking was observed among 26.8% of nurse auxiliaries, 26.3% of nurses, 16.7% of physiotherapists, 27.6% of health managers and 27% of doctors. Among the 3,659 respondents to a study at the Hospices Civils de Lyon, the smoking rate among paramedics (nurses, nursing auxiliaries, and health managers) was 25.6%. Among doctors, pharmacists and dentists, the proportion of smokers is 17.3%, while it reaches 46% among technical and logistics staff. The same survey also showed that paramedical students are three times more likely to be smokers than medical students, and that night staff are 1.5 times more likely to be smokers, given the same age.

In mental health establishments, smoking is prevalent among both patients and healthcare professionals. Investigators now know that smoking affects mood and sleep. It aggravates all pathologies (somatic and psychological) and predisposes people to more diabetes, chronic bronchitis, cardiovascular disease, cancer, etc. It interacts with many psychotropic and analgesic drugs. Smoking screening and cessation assistance have become a quality of care indicator in mental health institutions.

Investigators hypothesise that easier access to smoking cessation consultations in the workplace will improve uptake of this support and encourage smoker carers to change their smoking habits, and that experimenting with this support will increase smoker carers' confidence in their ability to manage their patients' smoking.

The issue of smoking in patients with psychiatric comorbidity is a major one. Smoking significantly reduces their life expectancy: an average of 25 years less, compared with 10 years for smokers without mental disorders. Cardiovascular disease and cancer are the leading causes of premature death. Smoking also affects their quality of life by increasing their metabolic risk (diabetes), reducing their respiratory capacity (chronic obstructive bronchitis) and increasing their risk of chronic disabling pain (arteritis of the lower limbs). Healthcare professionals are expected to play an active role in the fight against smoking and to act as role models for those receiving care, promoting appropriate lifestyles to maintain good health.

Smoking by health professionals does not appear to be more prevalent at the Centre Hospitalier Alpes-Isère than in the general population: 25.9% compared with 25.5%, but this is still significant and probably contributes to the erroneous representations of smoking in psychiatry.

Today, the recommendations of the Haute Autorité de Santé specify that psychological support and assistance are the basis of treatment. Nicotine substitutes supplement this support if the smoker shows signs of nicotine dependence. For smoker health professionals, the offer of smoking counselling in the workplace is likely to encourage them to use these aids and to succeed.

In previous studies, investigators found cessation rates at 12 months of 33% in an intensive intervention group (NST, intensive advice and outpatient telephone follow-up) compared with 20% in a control group (minimal advice) (RR = 1.7; 95% CI: 1.1 to 2.7).

In a study of hospital smoking clinics, 29.5% of patients (schizophrenic patients were excluded) maintained cessation at 1 year: female gender and prematurely interrupted follow-up were significantly associated with the risk of relapse at 1 year.

With regard to smoker healthcare professionals, a meta-analysis published in 2020 of ten studies (6 cohort studies and 4 clinical trials) measured a one-year cessation rate of 21% following the application of pharmacological or behavioural interventions. Hajek et al. showed in a randomised trial that the vaporiser could double the success rate at 1 year compared with treatment with nicotine replacement therapy alone, if accompanied by behavioural support.

Invesigators therefore believe it is possible to achieve a one-year cessation rate of 30% with workplace consultations combining support, nicotine replacement therapy and/or a vapour device where appropriate.

Doctors' smoking status and attitudes towards smoking are known to influence their enthusiasm for advising their patients against smoking.

As the Nagahapitye et al. study made clear: 'It is reasonable to assume that a healthcare professional who is not a smoker or is a former smoker will be more committed and more convincing in spreading messages about smoking and cessation. Health professionals smoking habits are therefore an important factor in the prevention of tobacco-related diseases.

The hypotheses of PSYTaB are :

* To improve cessation and reduction rates among smokers working in mental health,
* To improve the management of their patients' smoking and representations of smoking.

This study may also highlight benefits for the healthcare establishment and society, notably in terms of reduction in sick leave rates.

This study involves no risk for the subject.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Health professional
3. Daily smoker of at least 1 cigarette or joint per day and every day
4. Willingness to quit smoking
5. Patient physically able and willing to undertake a carbon monoxyde measurement
6. Patient affiliated to a social security scheme or beneficiary of such a scheme
7. Signature of informed consent

Exclusion Criteria:

1. Smoking via vaporizer exclusively
2. Occasional (i.e. not daily) smoker or exhaled carbon monoxyde at inclusion < 9 ppm
3. Resignation, transfer or end of employment contract during the study period (1 year)
4. Unable to undergo study follow-up for geographical, social or psychological reasons
5. Persons under legal protection or unable to express their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Evalue the effectiveness of a counseling consultation in the workplace among smoker health professionals. | At 12 month
  Cessation rate at 12 months: At the 12-month visit, no smoking in the last 7 days (self-reported) confirmed by a measurement of exhaled carbon monoxyde < 9 ppm.

SECONDARY OUTCOMES:
Prevalence of anxiety and depressive disorders | at inclusion
  Mean Hospital Anxiety and Depression Scale scores To screen for anxiety and depressive symptoms, the following interpretation can be proposed for each of the scores (A and D) Total Score [0;21]
  * 7 or less: no symptoms
  * 8 to 10: doubtful symptomatology
  * 11 or more: definite symptomatology
Prevalence of chronic pain | at inclusion
  Pain numerical scale > 3/10 for 3 months or more
Prevalence of chronic fatigue | at inclusion
  Pichot scale, cut-off = 22
Effectiveness of counseling consultation on anxiety and depressive disorders | at inclusion, 6 months and 12 months
  Mean Hospital Anxiety and Depression Scale scores To screen for anxiety and depressive symptoms, the following interpretation can be proposed for each of the scores (A and D), Total score [0;21]
  * 7 or less: no symptoms
  * 8 to 10: doubtful symptomatology
  * 11 or more: definite symptomatology
Effectiveness of counseling consultation on pain | at inclusion, 6 months and 12 months
  Mean Pain Numerical Scale in the last 24 hours. Numerical scale from 0 to 10. Note 0 corresponds to "no pain". Note 10 corresponds to "maximum imaginable pain".
Effectiveness of counseling consultation on chronic fatigue | at inclusion, 6 months and 12 months
  Pichot scale score Total Score [0; 32] A total > 22 indicates excessive fatigue
Effectiveness of counseling consultation on the sense of personal efficacy with consumption and management of patients' smoking habits | at inclusion , 12 months.
  Numerical scale from 0 to 10 (0 means 'I'm absolutely sure I won't make it' and 10 means 'I'm absolutely sure I'll make it')
Effectiveness of counseling consultation on use of ancillary products | at inclusion, 12 months
  Rate of subjects using ancillary products and search for other uses and intentions (cessation or reduction)
Medico-economic impact of counseling consultation | between inclusion and 12-month follow-up
  Number of sick leave days
Prevalence of burnouts | at inclusion
  Maslach scale score
  The questionnaire thus yields 3 scores:
  * Professional Exhaustion Score (SEP) Total Score [0;54] A SEP < 17 reflects a low degree of burnout. A SEP between 18 and 29 indicates a moderate degree of burnout. A SEP over 30 indicates a high degree of burnout (red zone).
  * Depersonalization/Loss of Empathy Score (SD) Total Score [0;30] An SD < 5 reflects a low degree of depersonalization. An SD between 6 and 11 indicates a moderate degree of depersonalization. An SD greater than 12 indicates a high degree of loss of empathy (red zone).
  * Personal Accomplishment Score (SAP). Total Score [0;48] A SAP < 33 reflects a low degree of personal fulfillment (red zone). An SAP between 34 and 39 reflects a moderate degree of personal fulfillment. An SAP above 40 indicates a high degree of personal fulfillment.
  If both SAP and SD scores are in the red, the risk of Burn-out is very high, especially if the degree of personal fulfillment is also in the red.
Determine the profile of the smoker health professionals | at inclusion
  Data collection: gender, age, profession; level of dependence (Fagerstrom score); level of motivation to smoke and to use cannabis, if applicable (Richmond scale); and level of confidence in managing their patients' tobacco dependence.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Jenny, Medical doctor, Study Chair — Hospital Center Alpes-Isère
Locations (1):
- Groupe Hospitalier Mutualiste Grenoble, Grenoble, isere, France

IPD SHARING:
Plan to Share IPD: No